CLINICAL TRIAL: NCT03217331
Title: CRD-102 for Right Heart Failure in Patients With Left Ventricular Assist Devices
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cardiora Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARD-LV01
Record Dates: First submitted 2017-07-05; First posted 2017-07-14 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Right Heart Failure; Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CRD-102 Treatment (Experimental): CRD102 Treatment
  Interventions: Drug: CRD-102

INTERVENTIONS:
Drug: CRD-102 — 14 mg CRD-102 capsules administered twice daily orally for 14 days.

SUMMARY:
This is a Phase 1b/IIa, single centre, non-randomised open-label uncontrolled study to assess safety, effect and PK of oral CRD-102 in patients with RHF associated with the presence of an LVAD.

DETAILED DESCRIPTION:
The study will be conducted over a 40 day time period inclusive of screening and follow up time periods. Eligible subjects will receive oral CRD-102 for 14 days.

ELIGIBILITY:
Inclusion Criteria:

Patients are enrolled only if they met the following criteria.

1. Males and females aged 18-85 years inclusive
2. Have received a LVAD (HeartWare HVAD, HeartMate II) at least 30 days prior to screening.
3. Stable LVAD patients with evidence of ongoing right heart failure as evidenced by raised right atrial pressure indicated by JVP >6cm OR measured right atrial pressure ≥12mmHg within the 3 months prior to or at Baseline OR dilated IVC on echocardiography PLUS all of the following;

   1. ongoing diuretic therapy;
   2. echocardiography in the 3 months prior to or at Baseline showing at least mild impairment in overall RV systolic function by visual assessment together with a TAPSE < 14mm.
4. Able to give written informed consent and agree to adhere to all protocol requirements.
5. All patients will be required to have an implanted cardiaoverter defibrillator. (ICD)

Exclusion Criteria:

1. Hemodynamically unstable patients.
2. Hypotension (MAP<60 or systolic BP <90 mmHg) at Screening or Baseline
3. Hypertension (MAP>95 or systolic BP >130 mmHg) at Screening or Baseline
4. Ventricular tachycardia or ventricular fibrillation in the past 30 days or poorly controlled atrial fibrillation (ventricular rate >120 bpm)
5. Concurrent participation in another investigational device study or prior participation in which a device was implanted and remains in place
6. Receipt of any investigational research agent within 30 days or 5 half-lives (whichever is longer) prior to Baseline.
7. Current treatment with intravenous inotropes or levosimendan, or treatment within the 2 weeks prior to Screening
8. Significant renal (eGFR<25 ml/min/1.73 sq m) or hepatic (bilirubin >3mg/dL) impairment or anemia (Hb <90g/dL) at Screening or Baseline.
9. Expected heart transplantation within the study period.
10. Pregnancy
11. History of allergic reaction to milrinone or any excipients in the study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Safety: Subject incidence of adverse events | 40 days
  Number of adverse events as a measure of safety and tolerability.

OTHER OUTCOMES:
Exploratory: Pulmonary artery pressures (mmHg). | 40 days
  Changes compared to baseline in Pulmonary artery pressures (mmHg)
Exploratory: Left ventricular ejection fraction (%) | 40 days
  Changes compared to baseline in left ventricular ejection fraction (%)
Exploratory: Quality of life (KCCQ questionnaire) | 40 days
  Changes compared to baseline in Quality of life (KCCQ questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: David Kaye, MD PhD, Study Chair — Cardiora Pty. Ltd.
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No